CLINICAL TRIAL: NCT03999463
Title: Sevoflurane Effect on Left Atrial Performance: A Transoesophageal Echocardiographic Study on Patients Undergoing Coronary Artery Bypasses Grafting
Brief Title: Sevoflurane Effect on Left Atrial Performance: A Transoesophageal Echocardiographic Study
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dr.Ibrahim Mamdouh Esmat, Assistant Professor of Anesthesia and Intensive Care Department, Faculty of Medicine, Ain- shams University, Cairo, Egypt., Ain Shams University
Other Study IDs: R 35 / 2019
Record Dates: First submitted 2019-06-23; First posted 2019-06-26 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The left atrial performance is affected by the preload as well as the afterload. The LA active pumping is increased by stretching of the LA but within limits, after which the active pumping declines. The LV stiffness acts as the LA afterload. Whenever the LV stiffness increases, the overall emptying fraction becomes more pumpdependent

DETAILED DESCRIPTION:
The echocardiographic assessment of the LA was frequently overlooked. While left atrial performance reflects both systolic and diastolic functions of the LV, it looks like more studies are being conducted to detect the effect of different interventions on the left atrial size and function. Other studies focus on the prognostic value and the ability to risk stratify different cohorts of patients, based on the early recognition of deranged LA performance.

Many studies were conducted on the effect of inhalational anesthetics on the left atrial function. Yet the results are inconclusive and sometimes contradictory. In a study on dogs, Gare Meir and his colleagues proved that desflurane, sevoflurane, and isoflurane depress left atrial contractility, delay relaxation, reduce chamber stiffness, preserve reservoir and conduit function, and impair left atrial-left ventricular coupling in vivo. Volatile anesthetics may cause impairment of both left atrial (LA) and left ventricular (LV) contractility. The mechanisms suggested were a decrease in the influx of calcium via voltage gated calcium channels as well as a decrease in calcium availability from sarcoplasmic reticulum.Echocardiographic assessment of the LA volumetric measures is comparable to that of Cardiovascular Magnetic Resonance (CMR) with clinically irrelevant difference. This makes echocardiographic assessment of LA volumes reliable, cheaperand easier to obtain.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ischemic heart disease
* Elective coronary artery bypass grafting.

Exclusion Criteria:

* Atrial or ventricular dysrhythmias,
* Associated mitral valve disease,
* Ejection Fraction <40%,
* Emergency coronary artery bypass grafting,
* Pericardial disease
* Contraindication to perform a TEE, e.g. Esophageal tumor

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients of any sex,40-75 years, maintaining sinus rhythm undergoing elective with preserved left ventricular systolic function.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
intraoperative transoesophageal echocardiography to test the effect of Sevoflurane on left atrial performance | 30 Minutes (Start point: After induction of anesthesia and before starting sevoflurane (first set of data). End point: After achieving one MAC sevoflurane anesthesia and before skin incision (second set of data)).
  Mitral inflow early diastolic velocity (meter/second)(m/s)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain-Shams University Hospitals, Cairo, Egypt